CLINICAL TRIAL: NCT01147965
Title: A Phase I/II Study of Active Immunotherapy With Ad5 [E1-,E2b-]-CEA(6D) Vaccine in Patients With Advanced or Metastatic Malignancies Expressing CEA
Brief Title: QUILT-3.038: Active Immunotherapy CEA Vaccine in Patients With Malignancies Expressing CEA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NantCell, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QUILT-3.038
Record Dates: First submitted 2010-06-15; First posted 2010-06-22 (Estimated); Results first posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer; Lung Cancer; Breast Cancer; Prostate Cancer
Keywords: Colon Cancer; Lung Cancer; Breast Cancer; CEA; Prostate Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Lung Neoplasms; Breast Neoplasms; Prostatic Neoplasms; Colonic Neoplasms | interventions — Ad5(E1-,E2b-)-CEA(6D) vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (Experimental): Cohort 1: Ad5 [E1-, E2b-]-CEA(6D) at a dose of 1 x 10^9 particles
  Interventions: Biological: Ad5 CEA Vaccine
- Cohort 2 (Experimental): Cohort 2: Ad5 [E1-, E2b-]-CEA(6D) at a dose of 1 x 10^10 particles
  Interventions: Biological: Ad5 CEA Vaccine
- Cohort 3 (Experimental): Cohort 3: Ad5 [E1-, E2b-]-CEA(6D) at a dose of 1 x 10^11 particles
  Interventions: Biological: Ad5 CEA Vaccine
- Cohort 4 (Experimental): Cohort 4 (Phase II Cohort at MTD): Ad5 [E1-, E2b-]-CEA(6D) at a dose of 1 x 10^11 particles
  Interventions: Biological: Ad5 CEA Vaccine
- Cohort 5 (Experimental): Cohort 5: Ad5 [E1-, E2b-]-CEA(6D) at a dose of 5 x 10^11 particles
  Interventions: Biological: Ad5 CEA Vaccine
- Cohort 6 (Experimental): Cohort 6: Ad5 [E1-, E2b-]-CEA(6D) at a dose of 5 x 10^11 particles
  Interventions: Biological: Ad5 CEA Vaccine

INTERVENTIONS:
Biological: Ad5 CEA Vaccine — Ad5 [E1-, E2b-]-CEA(6D) Vector Vaccine

SUMMARY:
The purpose of this study is to find out what effects (good and bad) that a cancer vaccine has on you and your cancer. The cancer vaccine is called Ad5 [E1-, E2b-]-CEA(6D)or ETBX-011 and is made by Etubics. This vaccine is based on a virus called an adenovirus but it has been changed to express the protein CEA that is found on some cancer cells. Therefore, the vaccine can tell the immune system to attack cancer cells which make CEA. The investigators are trying to determine whether giving this virus is safe and whether this causes a strong immune system attack on the cancer. ETBX-011 is an investigational drug.

DETAILED DESCRIPTION:
This is a phase I/II study with the primary purpose to determine the safety of immunization with Ad5 [E1-, E2B-]-CEA(6D), in patients with advanced or metastatic CEA-expressing malignancies. The secondary objectives are to evaluate CEA-specific immune responses to the immunizations and to obtain preliminary data on clinical response rate. The study population consists of patients with a histologically confirmed diagnosis of metastatic malignancy that is CEA positive who were previously treated with standard therapy known to have a possible survival benefit or refused such therapy. The study will determine the safety of three dosage levels of Ad5 [E1-, E2B-]-CEA(6D) vaccine (phase I component), and the maximally tolerated dose of Ad5 [E1-, E2B-]-CEA(6D) vaccine (phase II component). The study drug is Ad5 [E1-, E2B-]-CEA(6D) given by subcutaneous (SQ) injection every 3 weeks for 3 immunizations. We will evaluate safety in each cohort at least 3 weeks after the last patient in the previous cohort has received their first injection. A dosing scheme will be considered safe if <33% of patients treated at a dosage level experience DLT (e.g., 0 of 3, ≤1 of 6, ≤3 of 12 or ≤5 of 18 patients). We are currently enrolling up to 10 additional patients (Cohort 6) to evaluate safety, immunogenicity, and efficacy at the highest dose of vaccine.

ELIGIBILITY:
Inclusion Criteria

1. Histologically confirmed diagnosis of malignancy expressing CEA. Because this is a safety and immunogenicity study, patients are NOT required to have measurable or evaluable disease by Response Evaluation Criteria in Solid Tumors (RECIST).
2. For all tumor types other than colorectal, the tumor must express CEA as defined by immunohistochemical staining (at least 50% of the tumor with at least moderate intensity of staining) or a tumor known to be universally CEA positive (i.e. colon and rectal cancer). If colorectal cancer then, pathologic or clinical confirmation of adenocarcinoma is required.
3. Patients must have received treatment with standard therapy known to have a possible overall survival benefit.

   For the following common cancers, the following eligibility criteria apply:
   * Colorectal cancer: Must have received and progressed through at least one line of palliative chemotherapy consisting of one of the following regimens:

     * Palliative chemotherapy for metastatic colorectal cancer with 5 fluorouracil (or capecitabine) and oxaliplatin.
     * Palliative chemotherapy for metastatic colorectal cancer with 5 fluorouracil (or capecitabine) and irinotecan.
     * Palliative chemotherapy regimen for metastatic colorectal cancer that includes bevacizumab.
     * Colorectal cancer patients currently receiving palliative single-agent bevacizumab or cetuximab will be eligible for this trial and may continue these therapies concomitant with study treatment (if they have been on these single agent therapies for at least 3 months).
   * Breast cancer: Must have received and progressed through at least one line of chemotherapy for metastatic breast cancer consisting of one of the following regimens:

     * Palliative anthracycline- or taxane-based chemotherapy
     * Patients with tumors that over express HER2 (IHC 3+ or FISH+) must have received and progressed through at least one line of palliative therapy that combines trastuzumab with chemotherapy.
     * Breast cancer patients currently receiving palliative endocrine therapy or single-agent trastuzumab will be eligible for this trial and may continue these therapies concomitant with study treatment (if they have been on these single agent therapies for at least 3 months).
     * Patients who have been treated or offered the options of treatment with Bevacizumab (option clearly stated in the consent form).
     * Patients who have been treated or offered the options of treatment with Lapatinib (option clearly stated in the consent form).
   * Lung cancer: Must have received and progressed through chemotherapy for metastatic disease consisting of one of the following regimens:

     * Palliative platinum-based (cisplatin or carboplatin) chemotherapy if the patient has not received chemotherapy previously.
     * Palliative taxane-based (docetaxel or paclitaxel) or vinorelbine chemotherapy if the patient has received chemotherapy previously.
     * Lung cancer patients currently receiving palliative single-agent erlotinib or gefitinib will be eligible for this trial and may continue these therapies concomitant with study treatment (if they have been on these single agent therapies for at least 3 months).
   * Pancreatic cancer: Must have received and progressed through chemotherapy including gemcitabine.

     - Pancreatic cancer patients currently receiving palliative single-agent erlotinib will be eligible for this trial and may continue this therapy concomitant with study treatment (if they have been on this single agent therapy for at least 3 months).
   * For other malignancies, if a first line therapy with survival or palliative benefit exists, it should have been administered and there should have been progressive disease.
   * Patients who have received and progressed through first-line palliative chemotherapy must be advised regarding second-line therapy before being enrolled on this investigational study.
4. Karnofsky performance score of 70% or higher
5. Estimated life expectancy > 3 months
6. Age ≥ 21 years, but < 75
7. Adequate hematologic function, with WBC ≥ 3000/microliter, hemoglobin ≥ 9 g/dL (it is acceptable to have had prior transfusion), platelets ≥ 75,000/microliter; PT-INR <1.5, PTT <1.5X ULN
8. Adequate renal and hepatic function, with serum creatinine < 1.5 mg/dL, bilirubin < 1.5 mg/dL (except for Gilbert's syndrome which will allow bilirubin ≤ 2.0 mg/dL), ALT and AST ≤ 2.5 x upper limit of normal.
9. Patients who have received prior CEA-targeted immunotherapy are eligible for this trial, if this treatment was discontinued at least 3 months prior to enrollment.
10. Patients who are taking medications that do not have a known history of immunosuppression are eligible for this trial.
11. Ability to understand and provide signed informed consent that fulfills Institutional Review Board's guidelines.
12. Ability to return to the clinical site for adequate follow-up, as required by this protocol.

Exclusion Criteria

1. Patients with concurrent cytotoxic chemotherapy or radiation therapy should be excluded. There are no exclusions based on the number of prior chemotherapy, biologic, hormonal, or experimental regimens. Except for the permitted concomitant therapies (bevacizumab, cetuximab, trastuzumab, erlotinib, gefitinib, or hormonal therapy which patients must have been on for at least 3 months at the time of enrollment if they intend to continue them with the vaccine), there must be at least 3 months between any prior CEA-targeted immunotherapy and study treatment and at least 4 weeks between any other prior therapy (including radiotherapy) and study treatment. Patients must have recovered to grade 1 acute toxicities from prior treatment.
2. Patients with a history of or current brain metastases will not be permitted.
3. Patients with a history of autoimmune disease, such as but not restricted to, inflammatory bowel disease, systemic lupus erythematosus, ankylosing spondylitis, scleroderma, or multiple sclerosis. Autoimmune related thyroid disease and vitiligo are permitted.
4. Patients with serious intercurrent chronic or acute illness, such as cardiac disease (NYHA class III or IV), hepatic disease, or other illness considered by the Principal Investigator as unwarranted high risk for investigational drug treatment.
5. Patients with a medical or psychological impediment to probable compliance with the protocol should be excluded.
6. Concurrent (or within the last 5 years) second malignancy other than non melanoma skin cancer, cervical carcinoma in situ, controlled superficial bladder cancer, or other carcinoma in situ that has been treated.
7. Presence of an active acute or chronic infection including: a urinary tract infection, HIV (as determined by ELISA and confirmed by Western Blot). Patients with HIV are excluded based on immunosuppression, which may render them unable to respond to the vaccine; patients with chronic hepatitis are excluded because of concern that hepatitis could be exacerbated by the injections.
8. Patients on steroid therapy (or other immunosuppressives, such as azathioprine or cyclosporin A) are excluded on the basis of potential immune suppression. Patients must have had 6 weeks of discontinuation of any steroid therapy (except that used as pre-medication for chemotherapy or contrast-enhanced studies) prior to enrollment.
9. Pregnant and nursing women should be excluded from the protocol since this research may have unknown and harmful effects on an unborn child or on young children. If the patient is sexually active, the patient must agree to use a medically acceptable form of birth control while receiving treatment and for a period of 4 months following the last vaccination therapy. It is not known whether the treatment used in this study could affect the sperm and could potentially harm a child that may be fathered while on this study.
10. Patients with acute or chronic skin disorders that will interfere with injection into the skin of the extremities or subsequent assessment of potential skin reactions will be excluded.
11. Patients will be allowed warfarin 1mg po qd other than for port prophylaxis.
12. Patients with metastatic disease which is determined to be resectable will be excluded.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2010-07-16 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Duke Cancer Research Institute, Duke University, Durham, North Carolina
  - Medical Oncology Associates, PS, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Morse MA, Chaudhry A, Gabitzsch ES, Hobeika AC, Osada T, Clay TM, Amalfitano A, Burnett BK, Devi GR, Hsu DS, Xu Y, Balcaitis S, Dua R, Nguyen S, Balint JP Jr, Jones FR, Lyerly HK. Novel adenoviral vector induces T-cell responses despite anti-adenoviral neutralizing antibodies in colorectal cancer patients. Cancer Immunol Immunother. 2013 Aug;62(8):1293-301. doi: 10.1007/s00262-013-1400-3. Epub 2013 Apr 30. PMID 23624851
- [Result] Balint JP, Gabitzsch ES, Rice A, Latchman Y, Xu Y, Messerschmidt GL, Chaudhry A, Morse MA, Jones FR. Extended evaluation of a phase 1/2 trial on dosing, safety, immunogenicity, and overall survival after immunizations with an advanced-generation Ad5 [E1-, E2b-]-CEA(6D) vaccine in late-stage colorectal cancer. Cancer Immunol Immunother. 2015 Aug;64(8):977-87. doi: 10.1007/s00262-015-1706-4. Epub 2015 May 9. PMID 25956394

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Endpoints were tabulated as planned for the 43 patients by cohorts.
Groups:
- Cohort 1: 1x10^9 VP (0.5 mL)
- Cohort 2: 1x10^10 VP (0.5 mL)
- Cohort 3: 1x10^11 VP (0.5 mL)
- Cohort 4: Cohort 4 (Phase II): Ad5 [E1-, E2b-]-CEA(6D) at a dose of 1 x 10^11 particles
- Cohort 5: 5x10^11 VP (2.5 mL)
- Cohort 6: 5x10^11 VP (1.0 mL)
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Started | 3 | 4 | 7 | 14 | 6 | 9
Completed | 0 | 1 | 0 | 0 | 0 | 1
Not Completed | 3 | 3 | 7 | 14 | 6 | 8
Not completed — Progressive Disease | 3 | 3 | 5 | 9 | 5 | 5
Not completed — Death | 0 | 0 | 1 | 1 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Administration Of Alternative Therapy | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 4: (Phase II Cohort at MTD): Ad5 [E1-, E2b-]-CEA(6D) at a dose of 1 x 10^11 particles
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Total
Number analyzed (Participants) | 3 | 4 | 7 | 14 | 6 | 9 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (7.21) | 52.8 (7.80) | 54.0 (4.80) | 61.7 (8.31) | 55.5 (11.86) | 62.1 (7.46) | 58.8 (8.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 3 | 5 | 3 | 7 | 20
  Male | 2 | 3 | 4 | 9 | 3 | 2 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 0 | 0 | 1
  White | 3 | 4 | 7 | 11 | 6 | 9 | 40
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subjects with advanced or metastatic malignancies expressing CEA [Count of Participants; unit: Participants] | 3 | 4 | 7 | 14 | 6 | 9 | 43

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities
Description: The primary objective of this protocol is to determine the safety of immunization with Ad5 [E1-, E2b-]-CEA(6D) in patients with advanced or metastatic CEA-expressing malignancies. A dosing scheme will be considered safe if <33% of patients treated at a dosage level experience DLT (e.g., 0 of 3, ≤1 of 6, ≤3 of 12 or ≤5 of 18 patients).
Time Frame: Every 3 weeks for 9 weeks and every 3 months for 1 year
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 3 | 4 | 7 | 14 | 6 | 9
Participants | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Adverse Events
Time Frame: from the time of first dose to the 30 days past last dose of study drug, up to 330 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 3 | 4 | 7 | 14 | 6 | 9
Participants | 2 | 3 | 6 | 10 | 6 | 9

3. Secondary Outcome: Clinical Response Rate
Description: Clinical response was assessed for participants that achieve a clinical response of complete response (CR) or partial response (PR), according to RECISIT criteria (v1.0 for Cohorts 1-5 and v1.1 for Cohort 6). CR is defined as disappearance of all target lesions. PR is defined as >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: from first dose up to a year follow up
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 3 | 4 | 7 | 14 | 6 | 9
Participants | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Immune Response Against CEA - IFN-gamma Secreting Cells by Visit
Description: Cell mediated immune response was characterized using ELISpot assays performed on Peripheral Blood Mononuclear Cells to determine the number of IFN-gamma secreting cells.
Time Frame: Baseline (Week 0) up to Week 9
Measure: Mean (Standard Deviation); unit: Spot-forming cells per 1,000,000 PBMC
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 3 | 4 | 7 | 14 | 6 | 9
Spot-forming cells per 1,000,000 PBMC
  Baseline | 1.0 (1.73) | 8.5 (7.59) | 183.8 (448.83) | 32.8 (68.42) | 19.2 (32.88) | 29.5 (44.96)
  Week 3 | 6.7 (5.77) | 26.3 (43.04) | 270.4 (585.78) | 100.2 (154.91) | 181.3 (226.02) | 9.0 (18.73)
  Week 6 | 16.0 (23.52) | 1.7 (2.89) | 242.7 (449.40) | 78.7 (110.54) | 214.4 (191.11) | 27.6 (64.34)
  Week 9 | 0.0 (0.00) | 13.3 (23.09) | 59.0 (98.77) | 188.4 (364.15) | 82.4 (93.84) | 10.3 (13.29)

5. Secondary Outcome: CEA Antibody (ng/mL) by Visit
Description: Summary of CEA Antibody (ng/mL) by Visit
Time Frame: Baseline (Week 0) to Week 9
Population: Safety Population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 3 | 4 | 7 | 14 | 6 | 9
ng/mL
  Baseline | 0.0470 (0.02291) | 0.0310 (0.00400) | 0.0690 (0.09319) | 0.0709 (0.09117) | 0.3193 (0.21676) | 0 (0)
  Week 9 | 0.0760 (0.11953) | 0.0307 (0.01106) | 0.1157 (0.10571) | 0.0439 (0.05536) | 0.3665 (0.19723) | 0 (0)

ADVERSE EVENTS:
Time Frame: AE monitoring occurred from the time of informed consent to 30 days after the last dose of study drug, up to 330 days.
Description: Toxicity was graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
All-Cause Mortality (participants affected / at risk) | 3/3 | 3/4 | 6/7 | 8/14 | 4/6 | 7/9
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/4 | 2/7 | 1/14 | 1/6 | 2/9
Other Adverse Events (participants affected / at risk) | 2/3 | 3/4 | 6/7 | 10/14 | 6/6 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=4) | Cohort 3 (N=7) | Cohort 4 (N=14) | Cohort 5 (N=6) | Cohort 6 (N=9)
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=4) | Cohort 3 (N=7) | Cohort 4 (N=14) | Cohort 5 (N=6) | Cohort 6 (N=9)
Injection site reaction (General disorders) | 0 | 2 | 2 | 2 | 4 | 2
Fatigue (General disorders) | 0 | 1 | 0 | 2 | 3 | 4
Influenza like illness (General disorders) | 0 | 0 | 2 | 2 | 3 | 1
Pyrexia (General disorders) | 0 | 0 | 2 | 1 | 4 | 1
Chills (General disorders) | 0 | 0 | 1 | 2 | 2 | 1
Pain (General disorders) | 0 | 0 | 1 | 1 | 2 | 1
Injection site pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 2
Oedema (General disorders) | 0 | 0 | 2 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 2 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 2
Swelling (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Injection site induration (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Abdominal wall haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 3
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 2
Aspartate aminotransferase (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Biopsy skin (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Body temperature (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Menstruation normal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Protein total decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
White blood cell count (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chest wall mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Extrapyramidal disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 2 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Granuloma annulare (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Eyelid rash (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Swelling of eyelid (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Confidentiality Agreement in place.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-23): https://cdn.clinicaltrials.gov/large-docs/65/NCT01147965/Prot_SAP_000.pdf